CLINICAL TRIAL: NCT02188927
Title: Participation in Screening Colonoscopy in Response to an Advanced Notification Letter Plus Standard Invitation Versus Standard Invitation Only - a Population-based Randomized Controlled Trial
Brief Title: Effect of an Advanced Notification Letter on Screening Colonoscopy Participation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Collaborators: Centre of Postgraduate Medical Education (Other); European Union (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: TEAM/2012-9/5
Record Dates: First submitted 2014-07-11; First posted 2014-07-14 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Colorectal Cancer; Adenoma; Rectal Cancer
Keywords: Advanced notification letter; Standard invitation; Participation rate; Colonoscopy; Screening; Colorectal Neoplasms; Digestive System Diseases
MeSH Terms: conditions — Colorectal Neoplasms; Adenoma; Rectal Neoplasms; Digestive System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Implementation of ANL (Experimental): Intervention: Procedure : Implementation of routine Advanced Notification Letter included in Standard Invitation procedure
  Advanced Notification Letter will be implemented in invitation procedure and send two weeks before Standard Invitation (Standard Invitation will be send six weeks before planned screening colonoscopy)
  Interventions: Other: Implementation of ANL
- No included ANL (Active Comparator): Intervention: Behavioral : No included Advanced Notification Letter Sending Standard Invitation six weeks before planned screening colonoscopy
  Interventions: Behavioral: No included ANL

INTERVENTIONS:
Other: Implementation of ANL — Advance Notification Letter will be send two weeks before Standard Invitation for screening colonoscopy
  Arms: Implementation of ANL
Behavioral: No included ANL — Sending Standard Invitation only six weeks before planned screening colonoscopy
  Arms: No included ANL

SUMMARY:
Participation in a primary screening colonoscopy programs remains low. Advanced notification letter has been shown to increase participation in colorectal cancer screening with fecal occult blood testing and to be cost effective compared to standard invitation. It is unknown whether advanced notification letter increases participation rate in primary colonoscopy screening program.

We hypothesize that an Advance Notification Letter will have significant influence on participation in screening colonoscopy, comparing to standard invitation procedure and will thus result in higher efficiency of the program.

This randomized controlled study aims to compare the participation rate in screening colonoscopy in response to advanced notification plus standard invitation letter and standard invitation letter alone.

Material and methods: 6800 individuals aged 55-64 years will be drawn from the Population Registry and randomly assigned in a 1:1 ratio to the group invited for screening colonoscopy with advanced notification letter (send two weeks before standard invitation) plus standard invitation (send six weeks before planned screening colonoscopy) or to standard invitation only (send six weeks before planned screening colonoscopy). The sample size was calculated to detect 3% difference in participation rate between the groups (25% vs 28%) with 80% power.

ELIGIBILITY:
Inclusion Criteria:

* all individuals aged 55-64 years living in the counties covered with the organized CRC screening program and assigned to invitation to screening colonoscopy in the year 2014 are eligible for the study.

Exclusion Criteria:

* message from neighbor/family/post office on death of screenee (not updated in Population Registry)
* resident abroad (not updated in Population Registry)
* return of unopened letter of invitation and/or reminder (address unknown)
* diagnosis of CRC before the date of draw (not updated in the National Cancer Registry)

Ages: 55 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6800 (Estimated)
Dates: Start 2014-08; Primary Completion 2014-12 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Participation rate | three months after receiving invitation
  A percentage of invitees who undergo the screening colonoscopy. The sample size was calculated to detect 3% difference in participation rate between the groups (25% vs 28%) with 80% power.

SECONDARY OUTCOMES:
Response rate | three months after receiving invitation
  Estimation of the invitees' response rate to Standard Invitation and Advanced Notification Letter followed by Standard Invitation, before receiving Reminding Letter.

OTHER OUTCOMES:
Cost of including Advance Notification Letter | 1 year
  Total cost of including Advanced notification letter into the standard invitation procedure of this study group.

CONTACTS AND LOCATIONS:
Overall Officials: Karolina Janikowska, MD,MSc, Principal Investigator — The Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw, Poland; Jaroslaw Regula, MD, PhD, Study Chair — The Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw, Poland; Bartlomiej Kocot, Study Director — The Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw, Poland
Locations (1):
- The Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw, Poland, Warsaw, Mazovian, Poland